CLINICAL TRIAL: NCT02842515
Title: Study the Feasibility of Preparing an Autologous Advanced Therapy Medicinal Product for the Dental Pulp Regeneration in the Patient With Irreversible Pulp Inflammation or Dental Trauma
Brief Title: Feasibility of the Preparation of an Advanced Therapy Medicinal Product for Dental Pulp Regeneration
Acronym: Pulp'R
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: API/2014/47
Record Dates: First submitted 2016-07-18; First posted 2016-07-25 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Dental Stem Cells; Dental Pulp Regeneration

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Dental Pulp stem cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients requiring dental avulsion: Patients requiring dental avulsion
  Interventions: Other: teeth avulsion

INTERVENTIONS:
Other: teeth avulsion

SUMMARY:
Current endodontic treatment are based essentially on the ouster of parenchyma in case of trauma or irreversible pulp inflammation. These situations typically affect immature teeth in subjects aged from 8 to 15 years. Consequently, loss of a functional pulp is leads to discontinuation of root development and apical closure. The challenge for the clinician in the management of such situations is then preserving a pulp vitality. But current practices consist in a filling of the endo-canal system with an inert or semi-inert material. In this case, no pulp vitality is present. New treatment methods are needed. The objective Pulp'R is the study the feasibility of preparing an autologous combined advanced therapy medicinal product (ATMP) for dental pulp regeneration in the patient with irreversible pulp inflammation or dental trauma.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 8 to 15 years, with at least one tooth affected by a carious process,
* Patients aged from 8 to 15 years with major trauma preventing the maintenance of the tooth in the arch
* Patients aged from 16 to 20 years requiring avulsion germs wisdom teeth,
* Ability to carry out the extraction of pulp chamber content
* Signature of informed consent (from the patient and his guardian)
* Indication that the subject has understood the purpose and procedures required by the study and agrees to participate in the study and comply with the requirements and limitations inherent in this study,
* Patient with French social insurance.

Exclusion Criteria:

* Lack of ability to collect the dental pulp,
* Presence of necrosis in pulp complex or the possibility of preserving the pulp through appropriate techniques,
* Legal incapacity or limited legal capacity
* Patient unlikely to cooperate in the study and / or low cooperation anticipated by the investigator,
* Patient without health insurance,
* The patient is in the period of exclusion of another study,
* Patients with congenital pathology of dental pulp (amelogenesis and dentinogenesis imperfect)
* Patient with intrapulpal calcification or violations of pulp obliteration
* Teeth having external or internal inflammatory resorption
* Teeth diagnosed with pulp necrosis process
* Teeth undergoing fragmentation for their avulsion
* Time of pulp air exposition > 2 hours (risk of bacterial contamination)

Ages: 8 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Male or Female aged from 8 to 15 years, with at least one tooth affected by a carious process, or a major trauma preventing the maintenance of the tooth in the arch, or requiring avulsion germs wisdom teeth.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Number of stem cell lines established from pulp removed during either traumatic or carious teeth avulsion | 1 day